CLINICAL TRIAL: NCT00290498
Title: A Phase II Randomized Study of Rituximab-HCVAD Alternating With Rituximab-Methotrexate-Cytarabine Versus Standard Rituximab-CHOP Every 21 Days for Patients With Newly Diagnosed High Risk Aggressive B-Cell Non-Hodgkin's Lymphomas in Patients 60 Years Old or Younger
Brief Title: Study of Rituximab-HCVAD Alternating With Rituximab-Methotrexate-Cytarabine Versus Standard Rituximab-CHOP Every 21 Days for Patients With Newly Diagnosed High Risk Aggressive B-Cell Non-Hodgkin's Lymphomas in Patients 60 Years Old or Younger
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0054; NCI-2012-01355 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2006-02-10; First posted 2006-02-13 (Estimated); Results first posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Lymphoma
Keywords: Non-Hodgkin's Lymphoma; B-Cell Non-Hodgkin's Lymphoma; Lymphoma; Cyclophosphamide; Cytarabine; Doxorubicin; Hyper-CVAD; Methotrexate; Prednisone; Rituximab; Vincristine; R-CHOP; R-HCVAD; Dexamethasone; Decadron; Leucovorin; Ara-C; Cytosar; Cytoxan; DepoCyt; Cytosine arabinosine hydrochloride; AD; Hydroxydaunomycin hydrochloride; Neosar
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin; Lymphoma, B-Cell | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Dexamethasone; Calcium Dobesilate; Methotrexate; Cytarabine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): R-HCVAD + R-MTX/Ara-C ((Rituximab-HCVAD (rituximab, doxorubicin, cyclophosphamide, vincristine, and dexamethasone) alternating with Rituximab-Methotrexate-Cytarabine))
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Dexamethasone; Drug: Methotrexate
- Arm B (Active Comparator): R-CHOP ((Rituximab-CHOP (Rituximab, cyclophosphamide, vincristine, and prednisone))
  No longer recruiting for this study arm.
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Prednisone

INTERVENTIONS:
Drug: Rituximab — Arm A: Rituximab 375 mg/m² by vein on day 1, Cycle 1 and alternating cycles. Arm B: Rituximab 375 mg/m² on day 1, Cycle 2 and alternating cycles.
  Other Names: Rituxan
Drug: Cyclophosphamide — Arm A: Cyclophosphamide 300 mg/m^2 by vein (IVPB) over 3 hours every 12 hours x 6 doses on Days 2-4, Cycle 1 and alternating cycles.
  Arm B: Cyclophosphamide 750 mg/m² by vein day 1
  Other Names: Cytoxan; Neosar
Drug: Doxorubicin — Arm A: Doxorubicin 50 mg/m^2/day by vein over 15 minutes (12 hours after last dose of cyclophosphamide) on Day 5, Cycle 1 and alternating cycles.
  Other Names: AD; Hydroxydaunomycin hydrochloride
  Arms: Arm A
Drug: Vincristine — Arm A: Vincristine 1.4 mg/m^2 (maximum 2 mg) by vein (IVPB) on Days 5 (1-24 hours after last cyclophosphamide) and on day 12, Cycle 1 and alternating cycles.
  Arm B: Vincristine 1.4 mg/m^2 (maximum 2 mg) by vein (IVPB) on Days 5 (1-24 hours after last cyclophosphamide) and on day 12 of each cycle.
  Arms: Arm A
Drug: Dexamethasone — Arm A: Dexamethasone 40 mg by vein or by mouth daily x 4 on Days 2-5 and on days 12-15 of cycle 1 and alternating cycles.
  Other Names: Decadron
  Arms: Arm A
Drug: Methotrexate — Arm A: Methotrexate after finishing Rituximab, 200 mg/m2 by vein over 2 hours, then 800 mg/m2 by vein over 22 hours day 1 cycle 2.
  Arms: Arm A
Drug: Cytarabine — Arm B: Cytarabine 3 g/m^2 by vein over 2 hours every 12 hours X 4 doses on days 3 & 4, cycle 2 and alternating cycles.
  Other Names: Ara-C; Cytosar; DepoCyt; Cytosine arabinosine hydrochloride
  Arms: Arm B
Drug: Prednisone — Arm B: Prednisone 100 mg by mouth (as a pill, capsule, or tablet) once a day on Days 1-5, each cycle.
  Arms: Arm B

SUMMARY:
The overall goal of this clinical research study was to find out which of two different chemotherapy drug combinations, R-CHOP and R-HCVAD, is more effective in treating B-cell lymphoma.

At this point, all participants will now be assigned to the R-HCVAD arm of the study. Researchers will study the safety and effectiveness of this drug combination.

DETAILED DESCRIPTION:
This study originally involved 2 different study drug regimens, R-CHOP and R-HCVAD. R-CHOP is made up of rituximab, cyclophosphamide, vincristine, and prednisone, and is the most common treatment for patients with non-Hodgkin's lymphoma. This combination was compared with R-HCVAD, which is made up of rituximab, doxorubicin, cyclophosphamide, vincristine, and dexamethasone.

Rituximab (Rituxan®) is a humanized monoclonal antibody against cluster of differentiation antigen 20 (CD20) (a receptor in the surface of malignant B-cell lymphocytes). The drug has activity against aggressive and nonaggressive NHL of B-cell origin, and has been used in combination with chemotherapy. Cyclophosphamide is a type of drug know as an alkylating agent. Vincristine is a type of drug called vinca alkaloids. It is typically used in lymphomas, leukemias, and other tumors. Prednisone is a type of steroid. Dexamethasone is a steroid that may have activity against lymphomas. Methotrexate is an anti-cancer drug and a folic acid antagonist. It is used to treat solid tumors, lymphomas, leukemias, and autoimmune diseases.

When this study began, participants were randomly assigned (as in the flip of a coin) to 1 of 2 arms: Arm A (R-HCVAD alternating with a combination of rituximab, methotrexate, and Ara-C) or Arm B (R-CHOP). From this point on, all new participants will be treated with the Arm A combination, which has shown to be better.

If you are found to be eligible to take part in this study, you will be given the study drugs in 21-day cycles. The cycles will alternate between R-HCVAD and a combination of rituximab, methotrexate, and Ara-C. During Cycle 1 (the R-HCVAD cycle), you will receive rituximab through a needle in your vein (intravenously, or "IV"), on Day 1. The infusion will take about 1 hour. Cyclophosphamide will be given by IV every 12 hours for 3 days. Each infusion of cyclophosphamide will take about 3 hours. Doxorubicin will be given as a 15-minute infusion on Day 5 with the supervision of a nurse. Your doctor may also choose to give you the doxorubicin over 24-48 hours using a small pump that you will carry around your waist in a "fanny pack." You will not have to stay in the hospital to receive this study drug. Vincristine will be given by IV, on Days 5 and 12. Each vincristine infusion will take about an hour. Dexamethasone will be given by mouth (as a pill, capsule, or tablet) on Days 2-5 and 12-15. You will also be given other standard medications to help prevent possible side effects of these medications (such as nausea, vomiting, or rash).

In Cycle 2 (the rituximab-methotrexate-Ara-C cycle), you will receive rituximab on Day 1. You will receive methotrexate by IV (after finishing the rituximab) on Days 2 and 3. The infusion will take about 24 hours. You will be given a small "fanny pack" with a pump inside that will slowly infuse the drug. You do not have to stay in the hospital while the drug is being given. You will be given Ara-C every 12 hours on Days 3-4 (a total of 4 doses). You will be given other standard medications to help prevent possible side effects of these medications (such as nausea, vomiting, or rash) during this cycle also.

Leucovorin is given 12 hours after each methotrexate infusion. It is used to stop the action of the methotrexate and to prevent/lessen any side effects that the methotrexate may cause.

During treatment, you will have blood draws (between 2-3 tablespoons) every week for routine tests. Every 4 weeks during treatment , you will be asked questions about your medical history and have a physical exam to check for any side effects. Every 2 cycles (about every 8 weeks), you will have bone marrow biopsies performed (if they were positive before starting on this study), until they come back negative. You will have a positron emission tomography (PET) scan to see if the tumor is responding. Once the PET scan comes back negative, it will be up to your physician to decide if you need additional PET scan tests, and when. You will have CT scans of the chest, abdomen, pelvis, and neck every 2 cycles, if they were positive at the beginning of the study also. You may have additional testing done while on this study, if your physician feels that it is needed (for example, if it is needed to check for side effects).

You may receive additional medication called "CNS prophylaxis" before receiving the study treatments. Your doctor will discuss these medications with you. The "CNS prophylaxis" consists of an alternating dose of either doxorubicin or methotrexate. The methotrexate will be given either by IV pump or by a "lumbar puncture" (a needle inserted into the space between the vertebrae in your back to infuse the drug directly into the spinal area). The doxorubicin will be given by IV. Changes in the dose level of CNS prophylaxis will be approved if you are at risk for or are experiencing serious side effects.

You will receive the study drugs for up to 6-8 cycles on an outpatient basis. This means you will not have to be admitted to the hospital to receive the study drugs. You may be taken off study if the disease gets worse. If you experience intolerable side effects while taking any of the study drugs, your study doctor may decide to delay your treatment for up to 3 weeks (one study cycle) or to continue your therapy on the drugs at a lower dose. If the side effects become very severe, your doctor may decide to take you off of the study and stop the medication.

At the end of your scheduled treatments, you will be asked to return to the clinic for follow-up visits every 6 months for the first, second, third, and fourth year after treatment on this study. You will then be followed every year after that. If your doctor feels it is necessary, you may have blood tests (about 3-5 teaspoons) performed at these visits. You will have bone marrow biopsies every other year for the first 2 years, if they were positive before you started on this study, and then every year after that. At these visits, you will be asked about any side effects you may have experienced and whether or not your cancer has come back. If your doctor feels there is a chance that the cancer has come back, he or she may schedule x-rays or scans in order to check. You will also be asked about any other therapies you may be having to treat your cancer, if it has come back.

If you are taken off study for any reason, you will be asked to come back to the clinic for an end-of-treatment visit within 4 weeks from the last treatment. This visit will include a physical exam, routine blood tests (about 5-8 teaspoons), a blood-pregnancy test for women who are able to get pregnant, an ECG, and a chest x-ray.

This is an investigational study. All of the study drugs are approved by the FDA for the treatment of lymphoma. Up to 66 patients will take part in this study. All of the patients will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of previously untreated large B-cell Non Hodgkin's, Large Cell Lymphoma and B-Cell with high grade features. Other aggressive lymphomas such as Primary Mediastinal large B-cell Lymphomas will be also allowed to be included.
2. Patients with performance status of 0-2 (Zubrod Scale).
3. Serum bilirubin <1.5 mg/dl and serum creatinine < 2.0 mg/dl unless due to lymphoma; absolute neutrophil count (ANC) >1000/mm^3 and platelets >100,000/mm^3 unless due to lymphoma.
4. Cardiac ejection fraction 50% or greater.
5. Ages 16 - 60 years (due to the fact that CHOP-R is not studied enough in younger patients and is not considered standard of care).
6. Patients must be willing to receive transfusions of blood products.
7. Age adjusted International Prognostic Index Score of 2 or more
8. Previous steroids are allowed (if used to relieve some symptoms such as SVC, etc).

Exclusion Criteria:

1. Pregnancy (excluded due to the teratogenicity of the involved chemotherapy agents
2. Positive HIV serology because of poor tolerance to this intense chemotherapy regimen
3. Burkitt's lymphomas, and Mantle cell lymphoma, transformed follicular center cell lymphoma, follicular grade III.
4. Any clinical or cytological diagnosis of central nervous system (CNS) involvement
5. Any co-morbid medical, such as Child's Class C liver cirrhosis, end-stage renal disease, and symptomatic congestive heart failure, or psychiatric illnesses that preclude treatment with intense dose chemotherapy as determined by the primary investigator.
6. Concurrent or previous malignancy whose prognosis is poor (< 90% probability of survival at 5 years)
7. Active Hepatitis B or C. Chronic carriers for Hepatitis B will be excluded.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 67 (Actual)
Dates: Start 2005-08-01 (Actual); Primary Completion 2017-08-11 (Actual); Study Completion 2017-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luis E. Fayad, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient eligibility:>/16 -</60 years old and untreated Diffuse Large B-cell Lymphoma,stage II >/10cm mass or stage III/IV),Eastern Cooperative Oncology Group 0-2,age-adjusted Integrated Pulmonary Index of .2, and adequate organ function. Excluded:if they were pregnant,breast-feeding,or evidenced central nervous system lymphoma or active infections.
Pre-assignment Details: Three participants were screen failures. Eight participants were removed
Groups:
- R-HCVAD-MA: I.V. rituximab 375mg, cyclophosphamide 300mg, doxorubicin 50mg & vincristine 1.4mg - 2mg, & oral dexamethasone 40mg. Alternate R-MA: IV rituximab 375mg, methotrexate 200mg & 800mg 22h, & cytarabine 3g.
- R-CHOP: R-CHOP: Day 1 I.V. rituximab 375mg, cyclophosphamide 750mg, doxorubicin 50mg, vincristine 1.4mg max 2mg, and oral prednisone 100mg orally.
Period: Overall Study
Arm/Group | R-HCVAD-MA | R-CHOP
Started | 49 | 10
Completed | 41 | 10
Not Completed | 8 | 0
Not completed — Death | 2 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Ineligible | 3 | 0
Not completed — Non-Compliance | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- R-HCVAD/R-MA: I.V. rituximab 375mg, cyclophosphamide 300mg, doxorubicin 50mg & vincristine 1.4mg - 2mg, & oral dexamethasone 40mg. Alternate R-MA: IV rituximab 375mg, methotrexate 200mg & 800mg 22h, & cytarabine 3g.
- Total: Total of all reporting groups
Arm/Group | R-HCVAD/R-MA | R-CHOP | Total
Number analyzed (Participants) | 49 | 10 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 10 | 59
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (11) | 39 (11) | 42.5 (22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 5 | 20
  Male | 34 | 5 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 45 | 9 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 0 | 7
  White | 40 | 10 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 49 | 10 | 59

OUTCOME MEASURES:

1. Primary Outcome: Response Rate R-HCVAD vs. R-CHOP
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Groups:
- R-HCVAD: I.V. rituximab 375mg, cyclophosphamide 300mg, doxorubicin 50mg & vincristine 1.4mg - 2mg, & oral dexamethasone 40mg. Alternate R-MA: IV rituximab 375mg, methotrexate 200mg & 800mg 22h, & cytarabine 3g.
Arm/Group | R-HCVAD | R-CHOP
Number analyzed (Participants) | 49 | 10
Participants
  Complete Remission | 40 | 7
  Inevaluable | 2 | 1
  Progressive Disease | 1 | 1
  Partial Remission | 4 | 0
  Complete Remission Unconfirmed | 2 | 1

2. Secondary Outcome: Progression Free Survival (Rate)
Description: Progression free survival (PFS) for three years following therapy with Rituxan-HCVAD alternating with Rituximab with high -dose methotrexate/ara-C and standard R-CHOP in patients with newly diagnosed B-cell aggressive non-Hodgkin's lymphomas younger than 60 years old and with adjusted IPI 2 or higher adverse prognostic features.
Time Frame: 3 years post-therapy
Measure: Count of Participants; unit: Participants
Groups:
- R-HCVAD/MA: I.V. rituximab 375mg, cyclophosphamide 300mg, doxorubicin 50mg & vincristine 1.4mg - 2mg, & oral dexamethasone 40mg. Alternate R-MA: IV rituximab 375mg, methotrexate 200mg & 800mg 22h, & cytarabine 3g.
Arm/Group | R-HCVAD/MA | R-CHOP
Number analyzed (Participants) | 49 | 10
Participants | 35 | 7

ADVERSE EVENTS:
Time Frame: From the initiation of the regimen until the end of chemotherapy, an average of 3 years
Groups:
- RHCVAD: Rituximab 375mg/m2 intravenously on day 1,cyclophosphamide 300mg/m2 intravenously every 12 h for six doses on days 13,doxorubicin 50mg/m2 intravenously on day 5,vincristine 1.4mg/m2 or maximum 2mg intravenously on days 5 and 12,and dexamethasone 40mg intravenously or orally on days 25,alternating with RMA(cycles 2,4,6,)rituximab 375mg/2 intravenously on day 1,methotrexate 200mg/m2 over 2 h followed by 800mg/m2 over 22 h on day 1, and cytarabine 3g/m2 every 12 h for four doses on days 3 and 4, with a 21 day cycle.
- RCHOP: RCHOP consisted of rituximab 375mg/m2 intravenously on day 1,cyclophosphamide 750mg/m2 intravenously on day 1,doxorubicin 50mg/m2 intravenously on day 1 either over 15min or 48 h , vincristine 1.4mg/m2 or maximum 2mg intravenously,and prednisone 100mg orally on days 15,with a 21d cycle.
Arm/Group | RHCVAD | RCHOP
All-Cause Mortality (participants affected / at risk) | 4/49 | 0/10
Serious Adverse Events (participants affected / at risk) | 49/49 | 7/10
Other Adverse Events (participants affected / at risk) | 46/49 | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RHCVAD (N=49) | RCHOP (N=10)
ABDOMINAL CRAMPING (Gastrointestinal disorders) | 1 | 1
ALKALINE PHOSPHATASE INCR (Investigations) | 4 | 1
ALLERGIC REACTION DRUG (Immune system disorders) | 10 | 1
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 9 | 3
ALLERGY (OTHER) (Immune system disorders) | 1 | 1
ALOPECIA (Skin and subcutaneous tissue disorders) | 20 | 5
ALT,SGPT INCR (Investigations) | 17 | 3
ANOREXIA (Metabolism and nutrition disorders) | 1 | 1
AST,SGOT INCR (Investigations) | 17 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0
ATRIAL FLUTTER (Cardiac disorders) | 2 | 0
AUDITORY/EAR (OTHER) (Ear and labyrinth disorders) | 1 | 0
AUTOIMMUNE REACTION (Immune system disorders) | 1 | 0
BILIRUBIN INCREASE (Investigations) | 9 | 0
BLURRED VISION (Eye disorders) | 0 | 2
BLOOD BONE MARROW (OTHER) (Blood and lymphatic system disorders) | 1 | 0
BRUISING (NON-THROMBOPENIA) (Injury, poisoning and procedural complications) | 1 | 0
CANDIDIASIS (Infections and infestations) | 3 | 0
CHOLESTEROL,SERUM-HIGH (Investigations) | 1 | 0
COGNITIVE DISTURBANCE (Nervous system disorders) | 1 | 0
CONFUSION (Psychiatric disorders) | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 16 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 17 | 4
CREATININE INCREASE (Investigations) | 7 | 2
DEATH NOS (General disorders) | 2 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 2 | 0
DERMATOLOGY/SKIN (OTHER) (Skin and subcutaneous tissue disorders) | 1 | 0
DIABETES (Metabolism and nutrition disorders) | 3 | 0
DIARRHEA (Gastrointestinal disorders) | 11 | 2
DISTENSION/BLOATING (Gastrointestinal disorders) | 1 | 0
DIZZINESS (Nervous system disorders) | 14 | 3
DRUG FEVER (General disorders) | 1 | 0
DRY EYE (Eye disorders) | 2 | 0
DRY MOUTH (Gastrointestinal disorders) | 2 | 1
DRY SKIN (Skin and subcutaneous tissue disorders) | 3 | 0
DYSPHAGIA (Gastrointestinal disorders) | 2 | 0
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 22 | 3
DYSURIA (Renal and urinary disorders) | 1 | 1
EDEMA (General disorders) | 8 | 3
EDEMA:HEAD AND NECK (General disorders) | 2 | 0
EDEMA:LIMB (General disorders) | 13 | 3
EDEMA:TRUNK/GENITAL (General disorders) | 2 | 0
EDEMA (LARYNX) (General disorders) | 1 | 0
ELEV LDH (OTHER) (Investigations) | 6 | 3
ENDOCRINE (OTHER) (Endocrine disorders) | 1 | 0
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 5 | 0
FATIGUE (General disorders) | 31 | 2
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 27 | 2
FEVER UNKNOWN ORIGIN (General disorders) | 2 | 1
FEVER WITHOUT NEUTROPENI (General disorders) | 14 | 3
FLU-LIKE SYNDROME (General disorders) | 1 | 1
FLUSHING (Vascular disorders) | 4 | 0
GAIT/WALKING (General disorders) | 1 | 0
GASTRITIS (Gastrointestinal disorders) | 7 | 0
GERD (Gastrointestinal disorders) | 2 | 0
GASTROINTESTINAL (OTHER) (Gastrointestinal disorders) | 2 | 1
GRANULOCYTOPENIA (Investigations) | 0 | 1
HAND-FOOT SYNDROME (Skin and subcutaneous tissue disorders) | 4 | 0
HEADACHE (Nervous system disorders) | 1 | 0
HEARTBURN (Gastrointestinal disorders) | 5 | 0
HEMATOMA (Vascular disorders) | 0 | 1
HEMATURIA (Renal and urinary disorders) | 1 | 0
HEMOGLOBIN DECREASE (Investigations) | 48 | 7
HEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 1
HEMORRHAGE (Blood and lymphatic system disorders) | 8 | 1
HEMORRHOIDS (Gastrointestinal disorders) | 6 | 0
HORSENESS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
HOT FLASHES (Reproductive system and breast disorders) | 1 | 0
HYPERGLYCEMIA (Investigations) | 25 | 6
HYPERKALEMIA (Investigations) | 2 | 0
HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 1 | 0
HYPERTENSION (Cardiac disorders) | 9 | 0
HYPERTHYROIDISM (Endocrine disorders) | 1 | 0
HYPERURICEMIA (Investigations) | 4 | 5
HYPOALBUMINEMIA (Investigations) | 27 | 4
HYPOCALCEMIA (Investigations) | 15 | 4
HYPOGLYCEMIA (Investigations) | 1 | 1
HYPOKALEMIA (Investigations) | 15 | 4
HYPOMAGNESEMIA (Investigations) | 14 | 6
HYPONATREMIA (Investigations) | 7 | 2
HYPOPHOSPHATEMIA (Investigations) | 2 | 0
HYPOTENSION (Cardiac disorders) | 13 | 0
HYPOTHYROIDISM (Endocrine disorders) | 1 | 0
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 | 1
INFECTION(S) (Infections and infestations) | 47 | 6
INSOMNIA (Psychiatric disorders) | 12 | 2
LEUKOPENIA (Investigations) | 48 | 7
MEMORY IMPAIRMENT (Nervous system disorders) | 1 | 0
MENORRHAGIA (Reproductive system and breast disorders) | 1 | 0
METABOLIC/LABORATORY (OTHER) (Metabolism and nutrition disorders) | 1 | 1
MOOD ALTERATION (Psychiatric disorders) | 16 | 2
MUCOSITIS (Respiratory, thoracic and mediastinal disorders) | 20 | 3
MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 8 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 3 | 0
MYOSITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 30 | 6
NEUROPATHY:MOTOR (Nervous system disorders) | 1 | 3
NEUROPATHY:SENSORY (Nervous system disorders) | 20 | 4
NEUTROPENIA (Investigations) | 46 | 4
OBESITY (Metabolism and nutrition disorders) | 2 | 0
OBSTRUCTION,GI (Gastrointestinal disorders) | 2 | 0
OCULAR/VISUAL(OTHER) (Eye disorders) | 1 | 0
OLIGURIA (Investigations) | 1 | 0
PAIN (ABDOMEN NOS) (Gastrointestinal disorders) | 6 | 2
PAIN (ANUS) (Gastrointestinal disorders) | 0 | 1
PAIN (BACK) (Musculoskeletal and connective tissue disorders) | 10 | 1
PAIN (BONE) (Musculoskeletal and connective tissue disorders) | 5 | 1
PAIN (BREAST) (Reproductive system and breast disorders) | 1 | 0
PAIN (CHEST/THORAX) (Respiratory, thoracic and mediastinal disorders) | 7 | 0
PAIN (DENTAL/TEETH/PERID (General disorders) | 2 | 1
PAIN (EXTREMITY-LIMB) (Musculoskeletal and connective tissue disorders) | 6 | 0
PAIN (EYE) (Eye disorders) | 1 | 0
PAIN( HEAD/HEADACHE) (Nervous system disorders) | 22 | 3
PAIN (JOINT) (Musculoskeletal and connective tissue disorders) | 3 | 0
PAIN (MUSCLE) (Musculoskeletal and connective tissue disorders) | 7 | 2
PAIN (NECK) (Musculoskeletal and connective tissue disorders) | 5 | 0
PAIN (NEURALGIA/PERIPHERALNER (Nervous system disorders) | 1 | 0
PAIN (NOS) (General disorders) | 4 | 2
PAIN( ORALCAVITY) (Gastrointestinal disorders) | 1 | 0
PAIN (PELVIS) (Musculoskeletal and connective tissue disorders) | 1 | 0
PAIN (PLEURITIC) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PAIN( STOMACH) (Gastrointestinal disorders) | 1 | 0
PAIN (TESTICLE) (Reproductive system and breast disorders) | 2 | 0
PAIN (THROAT/PHARYNX/LARYNX) (Respiratory, thoracic and mediastinal disorders) | 3 | 0
PAIN (VAGINA) (Reproductive system and breast disorders) | 1 | 0
PALPITATIONS (Cardiac disorders) | 1 | 1
PERICARDIAL EFFUSION (Cardiac disorders) | 1 | 1
PETECHIAE (Blood and lymphatic system disorders) | 6 | 0
PHLEBITIS (Blood and lymphatic system disorders) | 1 | 0
PLATELETS DECREASED (Investigations) | 39 | 3
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 8 | 0
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 | 0
POLYURIA (Renal and urinary disorders) | 1 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 4 | 0
PRURITUS/ITCHING (Skin and subcutaneous tissue disorders) | 1 | 0
PULMONARY(OTHER) (Respiratory, thoracic and mediastinal disorders) | 1 | 1
PULMONARY EMBOLISM (Skin and subcutaneous tissue disorders) | 1 | 0
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 14 | 2
RENAL FAILURE (Renal and urinary disorders) | 4 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RHINORRHEA (Respiratory, thoracic and mediastinal disorders) | 6 | 0
RIGORS/CHILLS (General disorders) | 18 | 1
SENSORY (Nervous system disorders) | 2 | 1
SINUS BRADYCARDIA (Cardiac disorders) | 3 | 0
SINUS TACHYCARDIA (Cardiac disorders) | 9 | 0
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 1 | 0
STOMATITIS (Gastrointestinal disorders) | 3 | 2
SWEATING (Skin and subcutaneous tissue disorders) | 7 | 1
SYNCOPE (FAINTING) (Nervous system disorders) | 7 | 0
SYNDROMES (OTHER) (Vascular disorders) | 1 | 0
TACHYCARDIA (Cardiac disorders) | 2 | 1
TASTE ALTERATION (Gastrointestinal disorders) | 2 | 0
TEETH (Gastrointestinal disorders) | 2 | 0
THROMBOCYTOPENIA (Investigations) | 7 | 1
THROMBOSIS/THROMBUS/EMBOLISM (Vascular disorders) | 12 | 1
TINNITUS (Ear and labyrinth disorders) | 4 | 0
ULCERATION (Skin and subcutaneous tissue disorders) | 1 | 0
UPPER RESPIRATORY INFECT (Respiratory, thoracic and mediastinal disorders) | 1 | 0
URINARY FREQUENCY (Renal and urinary disorders) | 1 | 1
VAGINAL DRYNESS (Reproductive system and breast disorders) | 1 | 0
VASCULAR (OTHER) (Vascular disorders) | 1 | 1
VOICE CHANGES (Respiratory, thoracic and mediastinal disorders) | 3 | 1
VOMITING (Gastrointestinal disorders) | 24 | 5
WATERY EYE (Eye disorders) | 4 | 2
WEIGHT GAIN (Metabolism and nutrition disorders) | 1 | 1
WEIGHT LOSS (Metabolism and nutrition disorders) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RHCVAD (N=49) | RCHOP (N=10)
Neutrophils (Blood and lymphatic system disorders) | 46 | 4
Platelets (Blood and lymphatic system disorders) | 39 | 3
Febrile Neutropenia (Infections and infestations) | 25 | 2
Infection (Infections and infestations) | 33 | 5
Thrombosis/Embolism (Vascular disorders) | 12 | 1
Renal Failure (Renal and urinary disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-09-17): https://cdn.clinicaltrials.gov/large-docs/98/NCT00290498/Prot_SAP_000.pdf